CLINICAL TRIAL: NCT06403501
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Clinical Study to Evaluate the Efficacy and Safety of Clascoterone Cream 1% in Treatment of Subjects With Facial Acne Vulgaris
Brief Title: Efficacy and Safety of Clascoterone Cream 1% in Facial Acne Vulgaris
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Sunshine Mandi Pharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LWY23090C
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clascoterone Cream 1% (Experimental): Clascoterone Cream 1% (Winlevi)
  Interventions: Drug: Clascoterone
- Vehicle cream (Placebo Comparator): Vehicle cream manufactured to mimic look and feel of Clascoterone Cream 1% but without the active ingredient.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Clascoterone — Clascoterone Cream 1% (Winlevi) is indicated for the topical treatment of acne vulgaris in patients 12 years of age and older.
  Other Names: Winlevi (brand name)
  Arms: Clascoterone Cream 1%
Drug: Vehicle cream — Vehicle cream manufactured to mimic look and feel of Clascoterone Cream 1% but without the active ingredient.
  Arms: Vehicle cream

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of clascoterone cream, 1%, versus the vehicle cream applied twice daily for 12 weeks in subjects with facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with facial acne vulgaris (which includes the nose) from moderate to severe, has an Investigator's Global Assessment (IGA) score of 3 or 4; with at least 30 to a maximum of 75 inflammatory lesions (papules, pustules, and nodules) and 30 to a maximum of 100 non-inflammatory lesions (open and closed comedones);
* Male or female, 12 years of age or older;
* Subjects aged 18 years or older are required to provide informed consent and sign the written informed consent. A subject under 18 years of age must provide written informed assent and be accompanied by the parent or legal guardian at the time of consent signing.

Exclusion Criteria:

* Subject has greater than two (2) facial nodules;
* Subject has any skin pathology or condition that could interfere with the investigator's clinical evaluation of the investigational drug;
* Subject has used topical and systemic anti-acne medications or therapies;
* Subject has received hormonal therapy for acne treatment;
* Subject has used a skincare product with acne removal effect;
* Subject has other serious underlying diseases such as mental illness or malignant tumors;
* Subject has any of the clinically significant laboratory test indicators at screening;
* Subject has known hypersensitivity or previous allergic reaction to multiple drugs, or any of the active or inactive components of the test articles;
* Subject engaged in drug abuse or excessive alcohol intake;
* Subject has uncontrolled hypertension; Subject has poorly controlled diabetes;
* Subject is pregnant, lactating, or is planning to become pregnant during the study (both male and female); subject has positive pregnancy test result; subject is unable to practice highly effective contraception methods during the trial and within 3 months after the end of the trial;
* Subject is currently enrolled or was enrolled in other clinical trials within 3 months prior to the initiation of treatment;
* Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 692 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Success in Investigator's Global Assessment (IGA) | Week 12
  Percentage of subjects in each treatment group achieving "success" at Week 12, with "success" defined as an IGA score of "clear (score=0)" or "almost clear (score=1)" and at least a two-point reduction in IGA compared to Baseline.
Change From Baseline in Non-inflammatory Lesion (NIL) Counts | Week 12
  Absolute change from Baseline in non-inflammatory lesion counts in each treatment group at Week 12.
Change From Baseline in Inflammatory Lesion (IL) Counts | Week 12
  Absolute change from Baseline in inflammatory lesion counts in each treatment group at Week 12.

SECONDARY OUTCOMES:
Change From Baseline in Total Lesion Counts | Week 12
  Absolute change from Baseline in total lesions counts in each treatment group at Week 12.
Percent Change From Baseline in Total Lesion Counts | Week 12
  Percent change from Baseline in total lesions counts in each treatment group at Week 12.
Percent Change From Baseline in Inflammatory Lesion Counts | Week 12
  Percent change from Baseline in inflammatory lesions count in each treatment group at Week 12.
Percent Change From Baseline in Non-inflammatory Lesion Counts | Week 12
  Percent change from Baseline in non-inflammatory lesions count in each treatment group at Week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, China